CLINICAL TRIAL: NCT07064200
Title: Transversus Abdominis Plane (TAP) Blocks in Bariatric and General Surgery: Does Timing Matter?
Brief Title: TAP Block Timing Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 25-04028793
Record Dates: First submitted 2025-07-02; First posted 2025-07-14 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Bariatric or General Abdominal Surgeries; Bariatric Surgery Patients
Keywords: bariatric analgesia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Incision (Other): TAP block administration pre-incision
  Interventions: Other: TAP Block
- Post-Incision (Other): TAP block administration post-incision
  Interventions: Other: TAP Block

INTERVENTIONS:
Other: TAP Block — the TAP block is a regional anesthesia technique that targets the somatic nerves supplying the anterior abdominal wall.

SUMMARY:
This study investigates whether administering TAP blocks pre-incision provides superior postoperative pain control and reduces opioid use along with other medications compared to post-incision administration in patients undergoing elective abdominal surgeries.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 65 years
* Scheduled for elective bariatric surgery or other elective general abdominal surgeries
* Proficient in English sufficient to understand study procedures and communicate effectively
* Capable of providing informed consent

Exclusion Criteria:

* Individuals under 18 years of age (minors)
* Pregnant individuals
* Prisoners
* Individuals with cognitive impairments or otherwise unable to provide informed consent independently
* Individuals with known allergies or contraindications to local anesthetics used in TAP blocks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Mean change in opioid consumption (MME) from index procedure to 90 days post-op | Up to 90 days post-operatively
  Opioid dosage quantities will be measured in morphine milligram equivalents (MME)
Change in Pain Scores from index procedure on a numerical rating scale | 1, 3, 6, 24, 48, and 72 hours postoperatively
  Patient-reported pain on a scale of 1-10.

SECONDARY OUTCOMES:
1. Total Opioid Consumption in MME from Surgery to 90 Days Postoperatively | From end of surgery to 90 days post-op.
  Sum of all opioid use from surgery to 90 days, in MME
Patient Satisfaction Score with Postoperative Pain Management at Discharge | At hospital discharge (within 3-5 days post-op)
  Satisfaction score using a 5-point Likert scale survey before discharge.
Use of Non-Opioid Analgesics within 72 Hours | From end of surgery to 72 hours post-op
  Count of participants receiving non-opioid pain medications (e.g. acetaminophen, NSAIDs) within 72 hours post-op, including amount and type.
Number of Participants with TAP Block-Related Adverse Events | From TAP block administration to 90 days post-op.
  Incidence of adverse events (e.g. local anesthetic toxicity, infection, bleeding) related to TAP block.

CONTACTS AND LOCATIONS:
Overall Officials: Cheguevara Afaneh, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College - NewYork-Presbyterian Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices)
Supporting Information: Study Protocol
Time Frame: beginning at 9 months and ending 36 months following article publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee (:learned intermediary:) identifies for this purpose. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without the investigator support other than deposited metadata.